CLINICAL TRIAL: NCT06767683
Title: An Open-Label, Long-Term Extension Study to Investigate the Safety, Tolerability, and Durability of Treatment Effect of ALKS 2680 in Subjects With Narcolepsy Type 1 and Type 2 and Idiopathic Hypersomnia
Brief Title: A Long-Term Study of ALKS 2680 in Subjects With Narcolepsy and Idiopathic Hypersomnia
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALKS 2680-301
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Narcolepsy Type 1; Narcolepsy Type 2; Idiopathic Hypersomnia
Keywords: Narcolepsy; Narcolepsy Type 1; Narcolepsy Type 2; NT1; NT2; orexin-2 receptor agonist; sleep; sleep disorder; excessive daytime sleepiness; IH; Idiopathic Hypersomnia
MeSH Terms: conditions — Idiopathic Hypersomnia; Narcolepsy; Sleep Wake Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Narcolepsy Type 1 (NT1) (Experimental)
  Interventions: Drug: ALKS 2680, 4mg; Drug: ALKS 2680, 6mg; Drug: ALKS 2680, 8mg
- Narcolepsy Type 2 (NT2) (Experimental)
  Interventions: Drug: ALKS 2680, 10mg; Drug: ALKS 2680, 14mg; Drug: ALKS 2680, 18mg
- Idiopathic Hypersomnia (IH) (Experimental)
  Interventions: Drug: ALKS 2680, 10mg; Drug: ALKS 2680, 14mg; Drug: ALKS 2680, 18mg

INTERVENTIONS:
Drug: ALKS 2680, 4mg — Oral tablet containing 4 mg of ALKS 2680 for once daily administration
  Arms: Narcolepsy Type 1 (NT1)
Drug: ALKS 2680, 6mg — Oral tablet containing 6 mg of ALKS 2680 for once daily administration
  Arms: Narcolepsy Type 1 (NT1)
Drug: ALKS 2680, 8mg — Oral tablet containing 8 mg of ALKS 2680 for once daily administration
  Arms: Narcolepsy Type 1 (NT1)
Drug: ALKS 2680, 10mg — Oral tablet containing 10 mg of ALKS 2680 for once daily administration
  Arms: Idiopathic Hypersomnia (IH); Narcolepsy Type 2 (NT2)
Drug: ALKS 2680, 14mg — Oral tablet containing 14 mg of ALKS 2680 for once daily administration
  Arms: Idiopathic Hypersomnia (IH); Narcolepsy Type 2 (NT2)
Drug: ALKS 2680, 18mg — Oral tablet containing 18 mg of ALKS 2680 for once daily administration
  Arms: Idiopathic Hypersomnia (IH); Narcolepsy Type 2 (NT2)

SUMMARY:
The purpose of this study is to continue to measure the safety, tolerability, and durability of treatment effect in subjects with Narcolepsy Type 1 (NT1), Narcolepsy Type 2 (NT2), or Idiopathic Hypersomnia (IH) when taking ALKS 2680 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Was eligible for and has completed end of treatment visit of ALKS 2680 eligible parent study in NT1, NT2 or IH. The current eligible studies are ALKS 2680-201 (Vibrance-1), ALKS 2680-202 (Vibrance-2) and ALKS 2680-203 (Vibrance-3)
* Is willing and able, and in the opinion of the treating physician can safely discontinue any medications prescribed for the management of narcolepsy symptoms, as applicable, for 5 half-lives prior to Day 1 (for re-entry subjects), and for the duration of study (for all subjects)

Exclusion Criteria:

* Developed a new clinically significant health condition, ECG or laboratory abnormality, in the opinion of the Investigator or Sponsor, may impact the subject's participation in the study
* Is currently pregnant, breastfeeding, or planning to become pregnant during the study
* Is currently enrolled in another clinical study (other than the parent study) or used any investigational drug or device within 30 days prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Up to 100 Weeks

SECONDARY OUTCOMES:
Change in the mean sleep latency (MSL) on Maintenance of Wakefulness Test (MWT) | Baseline to Week 24
Change in Epworth Sleepiness Scale (ESS) | Baseline to 96 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alkermes, Inc.
Locations (43):
- United States (28):
  - Alkermes Investigator Site, Phoenix, Arizona
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Los Angeles, California
  - Alkermes Investigator Site, San Francisco, California
  - Alkermes Investigational Site, Stanford, California
  - Alkermes Investigational Site, Colorado Springs, Colorado
  - Alkermes Investigational Site, Brandon, Florida
  - Alkermes Investigational Site, Miami, Florida
  - Alkermes Investigational Site, Winter Park, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Macon, Georgia
  - Alkermes Investigational Site, Stockbridge, Georgia
  - Alkermes Investigational Site, Peoria, Illinois
  - Alkermes Investigational Site, Lansing, Michigan
  - Alkermes Investigational Site, Sterling Heights, Michigan
  - Alkermes Investigational Site, Lincoln, Nebraska
  - Alkermes Investigational Site, Middletown, New Jersey
  - Alkermes Investigational Site, Denver, North Carolina
  - Alkermes Investigational Site, Huntersville, North Carolina
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Dublin, Ohio
  - Alkermes Investigational Site, Abington, Pennsylvania
  - Alkermes Investigational Site, Wyomissing, Pennsylvania
  - Alkermes Investigational Site, Columbia, South Carolina
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, San Antonio, Texas
  - Alkermes Investigational Site, Sugar Land, Texas
- Australia (2):
  - Alkermes Investigational Site, Sydney, New South Wales
  - Alkermes Investigational Site, Bedford Park, South Australia
- Belgium (3):
  - Alkermes Investigational Site, Bruges, Brugge
  - Alkermes Investigational Site, Alken
  - Alkermes Investigational Site, Namur
- Alkermes Investigational Site, Prague, Czechia
- France (2):
  - Alkermes Investigational Site, Montpellier, Herault
  - Alkermes Investigational Site, Bordeaux
- Italy (3):
  - Alkermes Investigational Site, Bologna
  - Alkermes Investigational Site, Milan
  - Alkermes Investigational Site, Verona
- Alkermes Investigational Site, Zwolle, Netherlands
- Spain (3):
  - Alkermes Investigational Site, Madrid, Madrid
  - Alkermes Investigational Site, Barcelona
  - Alkermes Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided